CLINICAL TRIAL: NCT03041090
Title: Patterns and Prevalence of 18F-2-fluoro-2-deoxy-D-glucose (FDG) Extravasation in Positron Emission Tomography (PET)/ Computed Tomography (CT) Scans
Brief Title: Patterns and Prevalence of FDG Extravasation in PET/CT Scans
Acronym: Lucerno device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Lucerno Dynamics Limited Liability Company (LLC) (Unknown)
Responsible Party: Principal Investigator, Medhat M. Osman, MD., Sc.M., Ph.D., Professor of Radiology; Director of Nuclear Medicine & PET/CT, St. Louis University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SLU IRB # 26741
Record Dates: First submitted 2016-04-07; First posted 2017-02-02 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Intravenous Infiltration
Keywords: infiltration; extravasation; PET/CT; PET; PET-CT
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: All participants are included in the static imaging arm. Some participants were also included in the dynamic imaging arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Static Imaging participants (Experimental): This arm of the study assessed participants' static PET/CT images. These were the standard of care images acquired after their standard of care uptake time. These images were assessed visually by a board certified physician and using the Time Activity Curves from the sensor data.
  Intervention was Lucerno sensors (Lucerno Device Identity Document (LD ID), Lucerno Device 1 (LD1), Lucerno, Lara) placed on participant to monitor radiotracer activity at and around injection site.
  Interventions: Device: Lucerno ID (identification) System
- Dynamic image participants (Experimental): This arm of the study assessed participants' dynamic PET/CT images. These were the study related images of and around the injection site acquired during the participants' standard of care uptake time. These images were assessed visually by a board certified physician and using the Time Activity Curves from the sensor data.
  Intervention was Lucerno sensors (LD ID, LD1, Lucerno, Lara) placed on participant to monitor radiotracer activity at and around injection site.
  Interventions: Device: Lucerno ID (identification) System

INTERVENTIONS:
Device: Lucerno ID (identification) System — The Lucerno ID is intended to dynamically measure the uptake of radiotracer in a particular organ or body region during the radiotracer uptake period as part of nuclear medicine (NM) procedures. The Lucerno ID is indicated for use as a tool for trained healthcare professionals (technologists, NM physicians, and radiologists) to help assess whether a radiotracer injection has resulted in an infiltration. The LD ID can be used by healthcare professionals including nuclear medical technologists, nuclear medicine physicians, or any other medical staff in a NM facility, once they have received the necessary training into the use of the system.
  Other Names: LD ID (Lucerno Device identification), LD1 (Lucerno Device 1), Lucerno, Lara

SUMMARY:
PET (Positron Emission Tomography) images are used to help make patient management decisions in staging and treatment assessment, often after a cancer diagnosis.

Improper injections of PET tracers (dye) may occur approximately 15% of the time. This is known as extravasation or infiltration, and it compromises the doctor's ability to read the PET image. Often, the site where the tracer is injected into the vein (usually in the inside of the elbow) are not in the images taken, so reading physicians are unaware that an extravasation or infiltration has occurred.

Technology exists to capture time activity curves (amount of tracer in a location over a period of time) during the PET tracer uptake period (usually once the tracer is injected, the tracer circulates for 60 minutes prior to images), which can enable physicians to accurately detect extravasations and infiltration. This information is currently unavailable to physicians reading routine PET/CT (computed tomography) scans.

Time activity curves information gathered from these sensors during the circulation period appear to match the brief pictures taken approximately 70 minutes after the tracer injection.

This study will determine if these time activity curves correspond to PET images of the injection site taken during the tracer uptake period. If time activity curves correspond to PET images, they can be used to determine if the tracer was properly injected. If there was an improper injection, clinicians can be alerted to this fact and interpret the image with this additional information.

DETAILED DESCRIPTION:
PET (Positron Emission Tomography) images are used to help make patient management decisions in staging and treatment assessment, often after a cancer diagnosis.

Improper injections of PET tracers (dye) may occur approximately 15% of the time. This is known as extravasation or infiltration, and it compromises the doctor's ability to read the PET image. Often, the site where the tracer is injected into the vein (usually in the inside of the elbow) are not in the images taken, so reading physicians are unaware that an extravasation or infiltration has occurred.

Technology exists to capture time activity curves (amount of tracer in a location over a period of time) during the PET tracer uptake period (usually once the tracer is injected, the tracer circulates for 60 minutes prior to images), which can enable physicians to accurately detect extravasations. This information is currently unavailable to physicians reading routine PET/CT scans.

Time activity curves information gathered from these sensors during the circulation period appear to match the brief pictures taken approximately 70 minutes after the tracer injection.

This study will determine if these time activity curves correspond to PET images of the injection site taken during the tracer uptake period. If time activity curves correspond to PET images, they can be used to determine if the tracer was properly injected. If there was an improper injection, clinicians can be alerted to this fact and interpret the image with this additional information.

In oncology, whole-body PET/CT is typically performed from the head to the pelvic floor (eyes to thighs). The use of the term whole-body is misleading because the most commonly used field of view (FOV) for arms-up whole-body PET/CT protocols includes only the base of skull to the upper thighs and does not include the brain, skull, and large portions of both upper and lower extremities. In such FOV, the most commonly used site of injection, namely the antecubital fossa (inside of the elbow), is frequently not included in the imaging field. In the Frontiers in Oncology article, Osman also determined that based on the commonly used FOV at most PET/CT centers, that when infiltration is present, it may be unnoticed by clinicians in approximately 31% of the cases.

Lucerno Dynamics, a privately held company in North Carolina, has also discovered that the static image may be incapable of reporting on the quality of FDG administration during the ~60 minute uptake period. Lucerno's system has been used in two investigational studies at two centers. At one center, the system was used with 8 patients for a total of 15 scans. At the other center, the system was used with 40 patients for a total of 85 scans. Similar rates of infiltrations were found to those described in the published articles. Based on this experience, Lucerno has found that infiltrations can partially resolve during the uptake period, so that even if they are visible in the PET image, the image may not reveal the extent of the infiltration. This could severely and negatively impact research and therapy decisions and thus patient outcomes.

The Lucerno devices (Lucerno ID) are nonsignificant risk devices that add only 2-3 minutes to the current standard of care PET/CT scanning process. Lucerno ID sensors are applied to the patient's skin before the injection of the radiotracer and are removed after the FDG uptake period and prior to the PET/CT imaging process. The Lucerno ID has the ability to identify infiltrations, whether they are within or outside the FOV of reviewing clinicians, and can alert clinicians before their patient undergoes a compromised PET/CT scan due to the infiltration. This technology can prevent patients from receiving the additional CT radiation exposure of a compromised scan, can save cost, and can improve patient outcomes by ensuring more accurate PET scan interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18-90.
* Scheduled for a standard of care PET/CT scan at Sisters of Saint Mary (SSM) Saint Louis University (SLU) Hospital
* Willing to have self-adhesive sensors placed on the injections site, contralateral arm in approximately the same position as the injection site, liver, and over the subclavical area.
* If consenting to imaging during the PET/CT uptake period, the patient must be able to rest comfortably on the PET/CT scanning table for approximately 60 minutes during the circulation of the tracer for additional PET only imaging.

Exclusion Criteria:

* Persons (male or female) under age 18
* Persons with concerns about 4 adhesive sensors being placed on their bodies during the uptake period.
* Subjects unwilling to sign the consent document.
* Subjects who cannot consent for themselves
* Subjects who are not scheduled for a standard of care PET/CT exam at SLU hospital

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SSM Saint Louis University Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Coded data will be shared with our industry sponsor, Lucerno Dynamics

REFERENCES:
- [Result] Muzaffar R, Frye SA, McMunn A, Ryan K, Lattanze R, Osman MM. Novel Method to Detect and Characterize 18F-FDG Infiltration at the Injection Site: A Single-Institution Experience. J Nucl Med Technol. 2017 Dec;45(4):267-271. doi: 10.2967/jnmt.117.198408. Epub 2017 Nov 10. PMID 29127247
- [Result] Schaefferkoetter JD, Osman M, Townsend DW. The Importance of Quality Control for Clinical PET Imaging. J Nucl Med Technol. 2017 Dec;45(4):265-266. doi: 10.2967/jnmt.117.198465. Epub 2017 Oct 17. No abstract available. PMID 29042469
- [Derived] Lattanze RK, Osman MM, Ryan KA, Frye S, Townsend DW. Usefulness of Topically Applied Sensors to Assess the Quality of 18F-FDG Injections and Validation Against Dynamic Positron Emission Tomography (PET) Images. Front Med (Lausanne). 2018 Nov 1;5:303. doi: 10.3389/fmed.2018.00303. eCollection 2018. PMID 30443549
- See also: Published article: Novel Method to Detect and Characterize 18Fluoride-FDG Infiltration at the Injection Site: A Single-Institution Experience — https://www.ncbi.nlm.nih.gov/pubmed/29127247
- See also: Published article: The Importance of Quality Control for Clinical PET Imaging — https://www.ncbi.nlm.nih.gov/pubmed/29042469

RESULTS

PARTICIPANT FLOW:
Groups:
- Static Imaging Participants: This arm of the study assessed participants' static Positron Emission Tomography / Computed Tomography (PET/CT) images. These were the standard of care images acquired after their standard of care uptake time. These images were assessed visually by a board certified physician and using the Time Activity Curves from the sensor data. This arm also visually assessed the images at the injection site by a board certified physician.
- Dynamic Image Participants: This arm of the study assessed participants' dynamic Positron Emission Tomography / Computed Tomography (PET/CT) images. These were the study related images of and around the injection site acquired during the participants' standard of care uptake time. These images were assessed visually by a board certified physician and using the Time Activity Curves from the sensor data. This arm also visually assessed the images at the injection site by a board certified physician.
Period: Overall Study
Arm/Group | Static Imaging Participants | Dynamic Image Participants
Started | 109 | 24
Completed | 109 | 21 (3 consented subjects in the dynamic arm were not included in analysis due to technical errors.)
Not Completed | 0 | 3
Not completed — technical error | 0 | 3

BASELINE CHARACTERISTICS:
Population: Data were analyzed by physician review of the static standard of care PET/CT images and dynamic injection site images for visible evidence of radiotracer infiltration. The Time Activity Curves (TACs) generated from the applied sensors were independently assessed and the results compared to physician assessments of the PET/CT images.
Groups:
- Dynamic Arm: Participants that were already scheduled for a standard of care PET/CT study at a single institution could be included in this study. Those that chose to consent for this study had device sensors placed on the skin in four separate locations. The sensors could detect radiotracer near the injection site that was unavailable for circulation. During the 60 minute uptake, these subjects were scanned. After the 60 minute uptake period, the sensors were removed and participants continued with the normal PET/CT procedure. Participants also completed a questionnaire about the detector comfort. Dynamic arm (n=24 where 21 were analyzed) had 3 subjects that could not be analyzed due to technical errors, so 21 subjects were analyzed from this arm. Age and gender were not considered confounding factors and were not collected as part of the clinical study.
- Static Arm: Participants that were already scheduled for a standard of care PET/CT study at a single institution could be included in this study. Those that chose to consent for this study had device sensors placed on the skin in four separate locations. The sensors could detect radiotracer near the injection site that was unavailable for circulation. After the 60 minute uptake period, the sensors were removed and participants continued with the normal PET/CT procedure. Participants also completed a questionnaire about the detector comfort. The static arm included 109 subjects. Age and gender were not considered confounding factors and were not collected as part of the clinical study.
- Total: Total of all reporting groups
Arm/Group | Dynamic Arm | Static Arm | Total
Number analyzed (Participants) | 24 | 109 | 133
Age, Customized [Count of Participants; unit: Participants] — 18 to 90 years (adults only). Participant age was not collected as part of this clinical study as long as these participants were within the 18 to 90 year range. Population: Participant age was not included in analysis. The inclusion/exclusion criteria included that the subjects must be greater than or equal to 18 years and less than or equal to 90 years. Once the age was verified during the consent process, the specific age of the subject was not included in analysis.
Sex/Gender, Customized [Count of Participants; unit: Participants] — The genders included in this study were male and female. Participant gender was not collected as part of this clinical study. Population: Participant gender was not included in analysis. Al genders were included in the inclusion/exclusion criteria, so this data was not recorded nor included in analysis.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 109 | 133
Scheduled for a standard of care PET/CT [Count of Participants; unit: Participants] | 24 | 109 | 133

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Intraveneous Infiltration of FDG During Routine PET/CT Imaging by Visually Assessment of Interpreting Physicians
Description: Infiltrations of 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) during Positron Emission Tomography (PET) radiotracer administration can lead to sub-optimal images. We aim to compare rates of radiotracer presence near the injection site detected by physicians. Every subject that participates in an FDG-PET scan received an intervenous injection as part of this study. The number of participants by arm were provided in Static Imaging Participants and Dynamic Imaging Participants.
Time Frame: The time frame would be from the time the sensors were placed to the time the sensors were removed; no more than 2 hours.
Measure: Count of Participants; unit: Participants
Groups:
- Dynamic Arm: This arm includes the study participants that participated in dynamic image acquisition. Dynamic images include multiple static images over a specified amount of time per image.
- Static Arm: This arm includes the study participants that participated in static image acquisition.
Arm/Group | Dynamic Arm | Static Arm
Number analyzed (Participants) | 21 | 109
Participants | 17 | 32

2. Secondary Outcome: Number of Participants With Lucerno Sensor Device Detected Presence and/or Absence of Intravenous Infiltration
Description: Review collected Lucerno sensor graphical data. The Lucerno time activity curves will capture an amount of activity from the sensors and assess subjects for presence or absence of infiltration at injection site.
Time Frame: as for outcome 1
Population: The Time Activity Curve was studied that was provided from the sensor device among patients who underwent dynamic and static imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Dynamic Arm | Static Arm
Number analyzed (Participants) | 21 | 109
Participants | 14 | 26

3. Secondary Outcome: Percentage of Participants With Infiltrations Identified by Physicians and Sensor Device
Description: The percentage of participants with infiltrations identified by physicians compared with those identified by the Lucerno sensor device as a measure of agreement between the two methods.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Dynamic Arm | Static Arm
Number analyzed (Participants) | 21 | 109
percentage of participants | 66.67 | 23.85

ADVERSE EVENTS:
Time Frame: The time frame would be from the time the sensors were placed to the time it took the subjects to respond to questions; no more than 2 hours.
Description: Adverse events were collected during study participation. Participants completed a short questionnaire after participation to rate the pain of the sensor pads, pain of sensor placement, pain of sensor wires, and pain of removal of pads from skin.
Arm/Group | Dynamic Arm | Static Arm
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/109
Other Adverse Events (participants affected / at risk) | 0/24 | 0/109

LIMITATIONS AND CAVEATS:
Limitations: How the reading physicians visually assessed the radioactivity presence at the injection site may not consistently compare to the quantitative TACs. The motion of the patient during sensor measurement may affect measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03041090/ICF_000.pdf
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT03041090/Prot_001.pdf